CLINICAL TRIAL: NCT07402629
Title: Deep Learning-Based OCTA Quantification and Modeling for Predicting Long-Term Anti-VEGF Efficacy in mCNV
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1039
Record Dates: First submitted 2025-09-24; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Myopic Choroidal Neovascularization
Keywords: Deep learning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment-naïve patients with active mCNV at initial diagnosis, scheduled for intravitreal anti-VEGF
  Interventions: Other: No interventions beyond routine medical care

INTERVENTIONS:
Other: No interventions beyond routine medical care — No interventions beyond routine medical care

SUMMARY:
Myopic choroidal neovascularization (mCNV) is one of the sight-threatening complications secondary to pathological myopia. Intravitreal injection of anti-vascular endothelial growth factor (VEGF) is its first-line therapy. However, mCNV is prone to recurrence and long-term visual decline, and there is currently no definitive method for predicting long-term prognosis. This project aims to conduct a long-term follow-up and multi-dimensional quantitative analysis of mCNV using optical coherence tomography angiography (OCTA) images. It seeks to evaluate long-term prognostic indicators, such as recurrence and long-term visual acuity, following anti-VEGF therapy for mCNV, and to construct a deep learning (DL) prediction model for anti-VEGF efficacy based on multi-modal clinical data, ultimately enabling treatment personalization.

First, deep learning technology will be utilized to segment and quantitatively analyze mCNV in OCTA images, obtaining multi-dimensional quantitative parameters. These include OCTA-based The mCNV area and vessel junction(VJ). Patients will be followed up regularly for two years post-treatment, monitoring the number of injections, mCNV recurrence, OCT and OCTA quantitative parameters, fundus chorioretinal atrophy lesions, and visual acuity status. A multi-modal DL prediction model will be constructed, primarily based on the multi-dimensional quantitative characteristics of mCNV from OCTA images. This model will aim to identify sensitive indicators for predicting best-corrected visual acuity and recurrence after anti-VEGF therapy for mCNV and to clarify the relationship between therapeutic efficacy, baseline lesion status, and treatment regimen selection.

This research will open new avenues for clinically assessing the long-term efficacy of anti-VEGF therapy for mCNV, significantly improve the efficiency and accuracy of efficacy evaluation, and provide a critical reference for personalizing anti-VEGF treatment plans, holding substantial clinical significance.

ELIGIBILITY:
Inclusion Criteria:

* Myopic spherical equivalent greater than -6.0 diopters and/or axial length > 26.5 mm.
* Patients presenting with myopic fundus changes, as defined by the International Photographic Classification System for Myopic Maculopathy.
* Completion of a comprehensive ophthalmic examination at initial diagnosis, including Best Corrected Visual Acuity , slit-lamp examination, dilated fundus examination, intraocular pressure measurement, refractometry, axial length measurement, color fundus photography, Optical Coherence Tomography, OCT Angiography, and Fundus Fluorescein Angiography.
* Patients with active mCNV at initial diagnosis who are treatment-naïve.
* Final inclusion of all images required confirmation by two retinal specialists. Images with discrepant assessments were adjudicated by a senior researcher to reach a final decision.

Exclusion Criteria:

* Patients with choroidal neovascularization (CNV) due to causes other than myopia, such as age-related macular degeneration, adult-onset foveomacular vitelliform dystrophy, multifocal choroiditis, punctate inner choroidopathy, or retinoschisis.
* Poor-quality OCTA images, for example, those containing projection artifacts from overlying vessels at the mCNV lesion site, or excessively dark images dominated by thick outer choroidal vessels.
* Patients with a history of intraocular surgery, such as prior pars plana vitrectomy.
* Subjects who developed any of the above conditions during the follow-up period or who requested to withdraw from the study were removed from the experimental cohort.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with initially diagnosed, treatment-naïve active mCNV who are scheduled to undergo intravitreal anti-VEGF injection.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Best-Corrected Visual Acuity at 24 Months | Baseline to 24 months
  This outcome evaluates the change in best-corrected visual acuity (BCVA) from baseline to 24 months in eyes with myopic choroidal neovascularization receiving intravitreal anti-vascular endothelial growth factor treatment as part of routine clinical care. BCVA reflects functional visual outcome and is measured at each visit using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart under standardized testing conditions. BCVA values are recorded as ETDRS letter scores, and the primary assessment is the within-eye change from baseline to the 24-month follow-up visit.
Number of Recurrence Events During 24-Month Follow-up | Baseline to 24 months
  This outcome assesses disease activity by quantifying the number of recurrence events during the 24-month follow-up period in eyes with myopic choroidal neovascularization treated with intravitreal anti-vascular endothelial growth factor therapy. Recurrence is defined as the reappearance of active myopic choroidal neovascularization following an initial treatment response, as determined by clinical examination and imaging findings, including evidence of lesion activity that necessitates additional anti-vascular endothelial growth factor treatment.

SECONDARY OUTCOMES:
Change in Myopic Choroidal Neovascularization Area at 24 Months | Baseline to 24 months
  This outcome evaluates anatomical changes of the neovascular lesion by assessing the change in myopic choroidal neovascularization (mCNV) area from baseline to 24 months using optical coherence tomography angiography (OCTA). mCNV area is defined as the total en face area of the neovascular lesion identified on OCTA images. Measurements are obtained at baseline and follow-up visits to assess longitudinal changes in lesion size associated with anti-vascular endothelial growth factor treatment during the 24-month observation period.
Change In Number of Vessel Junctions at 24 Months | Baseline to 24 months
  This outcome assesses microvascular structural characteristics of the myopic choroidal neovascularization lesion by evaluating changes in the number of vessel junctions from baseline to 24 months using optical coherence tomography angiography (OCTA). Vessel junctions are defined as branching or connection points within the neovascular network visible on OCTA images. Changes in vessel junctions over time are used to describe morphological remodeling of the neovascular complex following intravitreal anti-vascular endothelial growth factor treatment during the follow-up period.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang HS, Kim JG, Kim JT, Joe SG. Prognostic factors of eyes with naive subfoveal myopic choroidal neovascularization after intravitreal bevacizumab. Am J Ophthalmol. 2013 Dec;156(6):1201-1210.e2. doi: 10.1016/j.ajo.2013.08.002. Epub 2013 Sep 25. PMID 24075429
- [Result] Wang Y, Hu Z, Zhu T, Su Z, Fang X, Lin J, Chen Z, Su Z, Ye P, Ma J, Zhang L, Li J, Feng L, Sun CB, Zhang Z, Shentu X. Optical Coherence Tomography Angiography-Based Quantitative Assessment of Morphologic Changes in Active Myopic Choroidal Neovascularization During Anti-vascular Endothelial Growth Factor Therapy. Front Med (Lausanne). 2021 May 7;8:657772. doi: 10.3389/fmed.2021.657772. eCollection 2021. PMID 34026789
- [Result] Hosoda Y, Miyata M, Uji A, Ooto S, Yamashiro K, Tamura H, Oishi A, Ueda-Arakawa N, Miyake M, Hata M, Muraoka Y, Takahashi A, Tsujikawa A. Novel Predictors of Visual Outcome in Anti-VEGF Therapy for Myopic Choroidal Neovascularization Derived Using OCT Angiography. Ophthalmol Retina. 2018 Nov;2(11):1118-1124. doi: 10.1016/j.oret.2018.04.011. Epub 2018 May 31. PMID 31047549
- [Result] Miyata M, Ooto S, Hata M, Yamashiro K, Tamura H, Akagi-Kurashige Y, Nakanishi H, Ueda-Arakawa N, Takahashi A, Kuroda Y, Wakazono T, Yoshikawa M, Yoshimura N. Detection of Myopic Choroidal Neovascularization Using Optical Coherence Tomography Angiography. Am J Ophthalmol. 2016 May;165:108-14. doi: 10.1016/j.ajo.2016.03.009. Epub 2016 Mar 10. PMID 26973049
- [Result] Rocholz R, Corvi F, Weichsel J, Schmidt S, Staurenghi G. OCT Angiography (OCTA) in Retinal Diagnostics. 2019 Aug 14. In: Bille JF, editor. High Resolution Imaging in Microscopy and Ophthalmology: New Frontiers in Biomedical Optics [Internet]. Cham (CH): Springer; 2019. Chapter 6. Available from http://www.ncbi.nlm.nih.gov/books/NBK554041/ PMID 32091844
- [Result] Li S, Sun L, Zhao X, Huang S, Luo X, Zhang A, Chen C, Wang Z, Liu C, Ding X. ASSESSING THE ACTIVITY OF MYOPIC CHOROIDAL NEOVASCULARIZATION: Comparison Between Optical Coherence Tomography Angiography and Dye Angiography. Retina. 2020 Sep;40(9):1757-1764. doi: 10.1097/IAE.0000000000002650. PMID 31652198
- [Result] Zhu Y, Zhang T, Xu G, Peng L. Anti-vascular endothelial growth factor for choroidal neovascularisation in people with pathological myopia. Cochrane Database Syst Rev. 2016 Dec 15;12(12):CD011160. doi: 10.1002/14651858.CD011160.pub2. PMID 27977064
- [Result] Soubrane G. Choroidal neovascularization in pathologic myopia: recent developments in diagnosis and treatment. Surv Ophthalmol. 2008 Mar-Apr;53(2):121-38. doi: 10.1016/j.survophthal.2007.12.004. PMID 18348878
- [Result] Wong TY, Ferreira A, Hughes R, Carter G, Mitchell P. Epidemiology and disease burden of pathologic myopia and myopic choroidal neovascularization: an evidence-based systematic review. Am J Ophthalmol. 2014 Jan;157(1):9-25.e12. doi: 10.1016/j.ajo.2013.08.010. Epub 2013 Oct 5. PMID 24099276
- [Result] Mi L, Zuo C, Zhang X, Liu B, Peng Y, Wen F. Fluorescein Leakage within Recent Subretinal Hemorrhage in Pathologic Myopia: Suggestive of CNV? J Ophthalmol. 2018 Aug 13;2018:4707832. doi: 10.1155/2018/4707832. eCollection 2018. PMID 30186627